CLINICAL TRIAL: NCT03458026
Title: Move Your Spondyl " Better Live Its Rheumatism With the Physical Activity "
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: LAMHNESS (Unknown); Azur sante (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-PP-12
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Spondyloarthritis
Keywords: activity; Connected object
MeSH Terms: conditions — Spondylarthritis; Motor Activity | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- connected object + SMS of physical activity reminders (Experimental): The patients will be included during their visit of follow-up and will receive a watch connected. They will have an information meeting for their to explain how step shows it. They will also receive advice to practise an adapted physical activity. During 12 weeks of SMS (text messages) every week to motivate them to realize these exercises.
  At the end of 12 weeks the connected watch will be deprived of them as well as SMS (text messages). They will have to realize an activity in autonomy during 12 weeks.
  At the end of the twenty-fourth week, they will get back their watch. They will have in more 1 session with a coach and 2 sessions to be made in autonomy during 12 weeks.
  In 36 week, they return the watch and finish the study.
  Interventions: Other: Connected object use combined with SMS (text messages) of physical activity reminders
- Without connected object (Other): The patients will be included during their visit of follow-up.They will have an information to practice suitable activity during 12 weeks At the end of 12 weeks, they realised follow-up. They will have to realize an activity in autonomy during 12 weeks.
  At the end of the twenty-fourth week, they will have 1 session with a coach and 2 sessions to be made in autonomy during 12 weeks.
  In 36 week, the study will be finished.
  Interventions: Other: Without connected object

INTERVENTIONS:
Other: Connected object use combined with SMS (text messages) of physical activity reminders — Watch connected used and receipt of SMS (text messages)
  Arms: connected object + SMS of physical activity reminders
Other: Without connected object — Any intervention except follow-up visit
  Arms: Without connected object

SUMMARY:
By this project, the investigators are going to try to demonstrate that to use objects connected to make a physical activity can have an impact on the clinical activity of the disease by bringing the subjects which present a spondyloarthritis to make a physical activity. The investigators shall show furthermore, than the use of connected objects also has better chances to glue the patients presenting a spondyloarthritis to a practice of regular physical activity that a simple recommendation.

DETAILED DESCRIPTION:
This project is aimed at subjects with Axial Spondyloarthritis and / or peripheral of the Alpes Maritimes and more specifically of the city of Nice and its surroundings. The subjects will be recruited by the hospital doctors (consultations, hospitalization). Patients will benefit from an inclusion visit in order to explain the protocol, sign the study consent and eliminate a possible contraindication to physical activity. Knowing that this is a physical activity adapted to the health of people and their physical abilities.

ELIGIBILITY:
Inclusion Criteria:

* Presenting a spondyloarthritis according to the criteria of the ASAS (l'Assessment of SpondyloArthritis international Society)
* Benefiting from a stable treatment by biotherapies for at least 3 months

Exclusion Criteria:

* Patient presenting a cardiac pathology should be decompensating
* Patients having a contraindication in the physical activity
* Lung affection making impossible the effort
* Patient already realizing a physical activity supervised in club or with sports coach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Number of pushes brought reported by the patient through a filled auto-questionnaire every week | After 12 weeks
  This questionnaire containing 3 items: did you present a push of your disease since the last filling of the questionnaire?,not, yes during 1 in 3 in the daytime,yes more than 3 days

SECONDARY OUTCOMES:
Moderators of the membership will be estimated thanks to the EMAPS (Scale of Motivation for Physical activity for health purposes) and thanks to the Big five | 12 weeks
  the EMAPS questionnaire will allow to quantify by the motivation of the patients to practice a physical activity.
  this questionnaire is specifically for health purposes.
The level of commitment in the physical activity will be estimated by the questionnaire GPAQ (Global Physical Activity Questionnaire) | 12 weeks
  the qestionnaire GPAQ is a scale to quantify overall physical activity (based on physical activity at work and in the home).
The function will be estimated by the BASFI (Bath Ankylosing Spondylitis Fonctional Index) | 12 weeks
The activity of the disease will be estimated by the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | 12 weeks
The activity of the disease will be estimated by the BASFI (Bath Ankylosing Spondylitis Fonctional Index) | 12 weeks
The activity of the disease will be estimated by the ASQOL (Ankylosing Spondylitis Quality of Life Questionnaire) | 12 weeks
  the ASQOL questionnaire is a quality of life scale. this questionnaire is specifically designed for patients with spondyloarthritis.
The activity of the disease will be estimated by the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | 24 weeks
The activity of the disease will be estimated by the BASFI (Bath Ankylosing Spondylitis Fonctional Index) | 24 weeks
The activity of the disease will be estimated by the ASQOL (Ankylosing Spondylitis Quality of Life Questionnaire) | 24 weeks
  the ASQOL questionnaire is a quality of life scale. this questionnaire is specifically designed for patients with spondyloarthritis.
The activity of the disease will be estimated by the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | 36 weeks
The activity of the disease will be estimated by the BASFI (Bath Ankylosing Spondylitis Fonctional Index) | 36 weeks
The activity of the disease will be estimated by the ASQOL (Ankylosing Spondylitis Quality of Life Questionnaire) | 36 weeks
  the ASQOL questionnaire is a quality of life scale. this questionnaire is specifically designed for patients with spondyloarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Background] Saraux A, Guillemin F, Guggenbuhl P, Roux CH, Fardellone P, Le Bihan E, Cantagrel A, Chary-Valckenaere I, Euller-Ziegler L, Flipo RM, Juvin R, Behier JM, Fautrel B, Masson C, Coste J. Prevalence of spondyloarthropathies in France: 2001. Ann Rheum Dis. 2005 Oct;64(10):1431-5. doi: 10.1136/ard.2004.029207. Epub 2005 Apr 7. PMID 15817661
- [Background] Passalent LA, Soever LJ, O'Shea FD, Inman RD. Exercise in ankylosing spondylitis: discrepancies between recommendations and reality. J Rheumatol. 2010 Apr;37(4):835-41. doi: 10.3899/jrheum.090655. Epub 2010 Mar 1. PMID 20194443
- [Background] Fongen C, Sveaas SH, Dagfinrud H. Barriers and Facilitators for Being Physically Active in Patients with Ankylosing Spondylitis: A Cross-sectional Comparative Study. Musculoskeletal Care. 2015 Jun;13(2):76-83. doi: 10.1002/msc.1088. Epub 2014 Nov 5. PMID 25370164
- [Background] O'Dwyer T, McGowan E, O'Shea F, Wilson F. Physical Activity and Exercise: Perspectives of Adults With Ankylosing Spondylitis. J Phys Act Health. 2016 May;13(5):504-13. doi: 10.1123/jpah.2015-0435. Epub 2015 Oct 28. PMID 26529384
- [Derived] Labat G, Hayotte M, Bailly L, Fabre R, Brocq O, Gerus P, Breuil V, Fournier-Mehouas M, Zory R, D'Arripe-Longueville F, Roux CH. Impact of a Wearable Activity Tracker on Disease Flares in Spondyloarthritis: A Randomized Controlled Trial. J Rheumatol. 2022 Oct;49(10):1109-1116. doi: 10.3899/jrheum.220140. Epub 2022 Jun 15. PMID 35705234